CLINICAL TRIAL: NCT03219788
Title: The Recovery Profile of Different Doses of Remifentanil After Desflurane Inhalational Anesthesia for Bariatric Surgeries: Two Centers Controlled Prospective Study
Brief Title: Remifentanil and Desflurane Inhalational Anesthesia in Bariatric Surgeries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr Mohamed Shaaban Ali, PhD, MD, Associate Profossor of Anesthesiology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00008715892
Record Dates: First submitted 2017-07-05; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia Emergence
Keywords: emergence; remifentanil; recovery; desflurene
MeSH Terms: interventions — Saline Solution; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1(Normal saline) (Placebo Comparator): Patients who will receive placebo (one ml normal saline). The drug will be given after closure of desflurane at an exhaled MAC of 0.3.
  Interventions: Drug: Normal Saline
- Group 2 (Remifentanil 0.1 ug/kg) (Active Comparator): Patients who will receive remifentanil at a dose of 0.1 ug/kg. The drug will be given after closure of desflurane at an exhaled MAC of 0.3.
  Interventions: Drug: Remifentanil 0.1 ug/kg
- Group 3 ((Remifentanil 0.2 ug/kg)) (Active Comparator): Patients who will receive remifentanil at a dose of 0.2 ug/kg. The drug will be given after closure of desflurane at an exhaled MAC of 0.3.
  Interventions: Drug: Remifentanil 0.2 ug/kg

INTERVENTIONS:
Drug: Normal Saline — All the patient will be anesthetized using a standard anesthetic technique. One ml normal saline will be given
  Other Names: Placebo
  Arms: Group 1(Normal saline)
Drug: Remifentanil 0.1 ug/kg — All the patient will be anesthetized using a standard anesthetic technique. One ml normal saline contains 0.1 ug/kg Remifentanil will be given
  Arms: Group 2 (Remifentanil 0.1 ug/kg)
Drug: Remifentanil 0.2 ug/kg — All the patient will be anesthetized using a standard anesthetic technique. One ml normal saline contains 0.2 ug/kg Remifentanil will be given
  Arms: Group 3 ((Remifentanil 0.2 ug/kg))

SUMMARY:
The number of obese and overweighted persons doubled since 1980. They are 600 million in 2014 all over the world. Obesity results in anatomical, physiological and pharmacological changes which represent a challenge for every anesthetist. Difficult airway increases by 30% with obesity and so awake extubation are the preferred technique. Coughing can be alleviated by opioid receptors which play a role in the cough reflex. Remifentanil may be useful as an ultra-short acting opioid and its effect swiftly and predictably disappears after cessation. An emergence cough is attenuated by remifentanil administered via continuous infusion (TCI), and the expected effective effect-site concentrations investigated have ranged from 1.5 to 2.5 ng.ml/L.

DETAILED DESCRIPTION:
The investigators designed this study to examine the effect of different small doses of Remifentanil on the incidence of cough reflex during emergence from anesthesia in obese patients undergoing bariatric surgery. The investigators will study if these small doses will delay the recovery of the patient or not. The other expected side effects will be observed eg. Respiratory depression. Time to the first painkiller required will be registered

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years
2. Subject has signed informed consent for bariatric laparoscopic surgery.
3. Subject must be ASA I or ASA II according to the American Society of Anesthetists classification.

Exclusion Criteria:

1. Age < 18 years.
2. Smoking patient.
3. Hypertension.
4. Bronchial asthma.
5. Obstructive sleep apnea syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in hemodynamic | within the first 24 hours
  Mean blood pressure and heart rate will be recorded before surgery and combined with all the other study items at the end of surgery, at the extubation time, after 5 minutes in PACU, after 10 minutes in Postanesthesia Care Unit (PACU) and he last registered reading in PACU.
antitussive effect | within the first 24 hours
  cough assessment at recovery time 0 no cough
  1. single cough
  2. cough episode less than five seconds or multiple coughs
  3. sustained attack of cough lasts more than five seconds

SECONDARY OUTCOMES:
Respiratory depression | within the first 24 hours
  In the postoperative period
Postoperative pain | within the first 24 hours
  The duration from extubation till the first painkiller and pain severity using VAS at the extubation time will recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Ali, MD, Principal Investigator — Associate profossor of anesthesiology